CLINICAL TRIAL: NCT01553149
Title: A Phase II Randomized Trial of Lenalidomide (NSC # 703813) in Pediatric Patients With Recurrent, Refractory or Progressive Juvenile Pilocytic Astrocytomas and Optic Pathway Gliomas
Brief Title: Low-Dose or High-Dose Lenalidomide in Treating Younger Patients With Recurrent, Refractory, or Progressive Pilocytic Astrocytoma or Optic Pathway Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00703; NCI-2012-00703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); s12-02726; COG-ACNS1022; ACNS1022; CDR0000728296; ACNS1022 (Other: Children's Oncology Group); ACNS1022 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2012-03-10; First posted 2012-03-14 (Estimated); Results first posted 2021-11-30 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Neurofibromatosis Type 1; Recurrent Childhood Pilocytic Astrocytoma; Recurrent Childhood Visual Pathway Glioma
MeSH Terms: conditions — Neurofibromatosis 1; Astrocytoma; Optic Nerve Glioma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (low-dose lenalidomide) (Experimental): Patients receive low-dose lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Other: Pharmacological Study
- Arm II (high-dose lenalidomide) (Experimental): Patients receive high-dose lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Other: Pharmacological Study

INTERVENTIONS:
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial studies how well low-dose lenalidomide works compared with high-dose lenalidomide in treating younger patients with juvenile pilocytic astrocytomas or optic nerve pathway gliomas that have come back (recurrent), have not responded to treatment (refractory), or are growing, spreading, or getting worse (progressive). Lenalidomide is classified as an immunomodulatory drug as it boosts the immune system. It has other potential anti-tumor effects, for example, it may stop the growth of tumor cells by blocking blood flow to the tumor. It is not yet known whether low-dose lenalidomide is more or less effective than high-dose lenalidomide in treating patients with juvenile pilocytic astrocytomas or optic nerve pathway gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the objective response rate in children with recurrent, refractory, or progressive juvenile pilocytic astrocytomas and optic pathway gliomas who are treated with Regimen A low-dose (20 mg/m^2/dose) or Regimen B high-dose (115 mg/m^2/dose) lenalidomide.

SECONDARY OBJECTIVES:

I. To estimate the event-free survival (EFS) (based on standard two-dimensional tumor measurements, determined by each institution) of children with recurrent, refractory, or progressive juvenile pilocytic astrocytomas and optic pathway gliomas who are treated with lenalidomide.

II. To compare response categories and EFS across the 3 magnetic resonance (MR) sequences (T2-weighted, fluid attenuated inversion recovery [FLAIR], T1-weighted post-contrast).

III. To correlate steady-state pharmacokinetics of lenalidomide (1 sample obtained between days 5-21) with objective response and EFS.

IV. To evaluate toxicities of long-term lenalidomide use.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I (Regimen A): Patients receive low-dose lenalidomide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

ARM II (Regimen B): Patients receive high-dose lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up annually for approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a body surface area (BSA) >= 0.4 m^2 at the time of study enrollment
* Patients must have a pilocytic astrocytoma or optic pathway glioma that has relapsed, progressed, or become refractory to conventional therapy; patients with neurofibromatosis (NF-1) are eligible
* Patients must have histologic verification of malignancy; histologic confirmation for patients with optic pathway gliomas will not be required
* Patients must have measurable residual disease, defined as tumor that is measurable in two perpendicular diameters on magnetic resonance imaging (MRI); for a lesion to be considered measurable, it must be at least twice the slice thickness on MRI (i.e. visible on more than one slice)
* To document the degree of residual tumor, the following must be obtained:

  * All patients must have a brain MRI with and without contrast (gadolinium) within 1 week prior to study enrollment; for patients on steroids, baseline MRI scans must be performed after at least 1 week at a stable or decreasing dose of steroids
  * All patients with a history of spinal or leptomeningeal disease, and those patients with symptoms suspicious of spinal disease, must have a spine MRI with and without contrast (gadolinium) performed within 2 weeks prior to study enrollment
* Patients must have a Lansky or Karnofsky performance status score of >= 60%; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have been treated with at least one prior treatment regimen that included carboplatin; patients who have received prior radiation therapy for this tumor are eligible
* Patients must have recovered (to Common Toxicity Criteria [CTC] version [v.]4.0 =< grade 1 unless indicated below) from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study, with the exception of alopecia, weight changes and grade I or II lymphopenia

  * Myelosuppressive chemotherapy: must not have received within 3 weeks of entry onto this study (6 weeks if prior nitrosourea or mitomycin-C)
  * Biologic (anti-neoplastic agent): at least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur
  * Immunotherapy: at least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
  * Monoclonal antibodies: at least 3 half-lives of the antibody after the last dose of a monoclonal antibody
  * Radiation therapy (RT): patients must have had their last fraction of craniospinal RT >= 6 months prior to study entry and their last fraction of focal RT >= 4 weeks prior to study entry; if the lesion used for on-study criteria is in the radiation field, there must be evidence of tumor progression after radiation therapy was completed
  * Study specific limitations on prior therapy:

    * Patients who have received thalidomide are eligible if all acute thalidomide-related toxicity has resolved
    * Patients must not have received lenalidomide previously
* Growth factor(s): must not have received within 2 weeks of entry onto this study
* Steroids: patients who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to baseline MRI
* Peripheral absolute neutrophil count (ANC) >= 1,000/uL
* Platelet count >= 100,000/uL (transfusion independent)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/m^2 OR a serum creatinine based on age/gender as follows:

  * 0.4 mg/dL (1 month to < 6 months of age)
  * 0.5 mg/dL (6 months to < 1 year of age)
  * 0.6 mg/dL (1 to < 2 years of age)
  * 0.8 mg/dL (2 to < 6 years of age)
  * 1.0 mg/dL (6 to 10 years of age)
  * 1.2 mg/dL (10 to < 13 years of age)
  * 1.5 mg/dL (male) or 1.4 mg/dL (female) (13 to < 16 years of age)
  * 1.7 mg/dL (male) or 1.4 mg/dL (female) (>= 16 years of age)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 110 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* No evidence of dyspnea at rest and a pulse oximetry > 94% if there is clinical indication for determination
* Patients must be able to swallow intact capsules
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Exclusion Criteria:

* Female patients who are pregnant are not eligible
* Lactating females are not eligible unless they have agreed not to breastfeed their infants while receiving protocol therapy and for 28 days after the last dose of lenalidomide
* Female patients of childbearing potential are not eligible unless they commit to complete abstinence or have been on 2 methods of birth control, including 1 highly effective method and 1 additional method at the same time (unless committing to complete abstinence of heterosexual intercourse) at least 28 days (4 weeks) prior to study enrollment; sexually active females must also agree to remain on 2 methods of birth control, during treatment (including during dose interruptions), and continuing for at least 28 days after the completion of protocol therapy; examples of methods of contraception are as follows:

  * Highly effective methods (must use at least 1):

    * Intrauterine device (IUD)
    * Hormonal (prescription birth control pills, injections, implants)
    * Tubal ligation
    * Partner's vasectomy
  * Additional effective methods:

    * Male condom
    * Diaphragm
    * Cervical cap The two methods of birth control requirement applies to all sexually active females unless they have undergone a hysterectomy or bilateral oophorectomy
* Female patients of childbearing potential (including those who commit to complete abstinence) are not eligible unless they agree to ongoing pregnancy testing and counseling every 28 days about pregnancy precautions and risks of fetal exposure
* Male patients of child fathering potential are not eligible unless they have agreed to use latex condoms during intercourse with a woman of childbearing potential while receiving treatment and for 28 days thereafter
* Patients with a history of thromboembolism unrelated to a central line, or patients with a known predisposition syndrome for thromboembolism are not eligible
* Patients who have an uncontrolled or untreated infection are not eligible
* Patients with known overt cardiac disease, including but not limited to a history of myocardial infarction, severe or unstable angina, clinically significant peripheral vascular disease, grade 2 or greater heart failure, or serious and inadequately controlled cardiac arrhythmia are not eligible
* Patients with a significant systemic illness that is not well-controlled in the opinion of the treating physician are not eligible

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2012-07-05 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine E Warren, Principal Investigator — Children's Oncology Group
Locations (126):
- United States (113):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Columbia Regional, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (5):
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Children's Hospital-Brisbane, Herston, Queensland
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (6):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Warren KE, Vezina G, Krailo M, Springer L, Buxton A, Peer CJ, Figg WD, William-Hughes C, Kessel S, Fouladi M, Gajjar A, Bowers D. Phase II Randomized Trial of Lenalidomide in Children With Pilocytic Astrocytomas and Optic Pathway Gliomas: A Report From the Children's Oncology Group. J Clin Oncol. 2023 Jun 20;41(18):3374-3383. doi: 10.1200/JCO.22.01777. Epub 2023 May 1. PMID 37126770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Started | 37 | 38
Completed | 32 | 18
Not Completed | 5 | 20
Not completed — Adverse Event | 0 | 9
Not completed — Physician Decision | 5 | 10
Not completed — Ineligible | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide) | Total
Number analyzed (Participants) | 37 | 38 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 37 | 38 | 75
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 8 [4 to 18] | 9 [2 to 17] | 9 [2 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 20 | 24 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 32 | 35 | 67
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 31 | 31 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 29 | 29 | 58
  Australia | 4 | 6 | 10
  Canada | 4 | 2 | 6
  New Zealand | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Demonstrate Complete or Partial Response
Description: Number of patients who demonstrate a complete or partial response as defined below:
  Complete Response - Complete disappearance of all known disease for at least 4 weeks;
  Partial Response - A reduction of at least 50% in the size of all measurable tumor as quantitated by the sum of the products of the largest diameters of measurable lesions when compared with that measurement at the time of study enrollment and maintained for at least 4 weeks.
Time Frame: 26 cycles of chemotherapy - up to 3 years after enrollment
Population: Only eligible patients are considered in the analysis of this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 37 | 37
Participants | 4 | 4

2. Primary Outcome: Number of Patients Who Demonstrate Early Progression
Description: Number of patients with disease progression during the first six months of protocol therapy. Disease progression is defined as ≥ 25% increase in the sum of the products of the largest diameters of the measurable lesions or the appearance of one or more new lesions when compared with the measurements of lesions at the time of enrollment.
Time Frame: Up to 180 days after enrollment
Population: Only eligible patients are considered in the analysis of this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 37 | 37
Participants | 6 | 4

3. Secondary Outcome: Event-free Survival [EFS]
Description: Estimated 3-year EFS where EFS is calculated as the time from study enrollment to disease progression, disease relapse, occurrence of a second malignant neoplasm, death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients without an event are censored at last contact.
Time Frame: Up to 3 years after study enrollment
Population: Only eligible patients are considered in the analysis of this outcome measure
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 37 | 37
Percent Probability | 37.84 [22.62 to 52.97] | 39.41 [23.72 to 54.74]

4. Secondary Outcome: Overall Survival [OS]
Description: Estimated 3-year overall survival is calculated as the time from study enrollment to death from any cause or last follow-up whichever occurs first. Kaplan-Meier method is used for estimation. Patients alive at last contact are censored at that time.
Time Frame: Up to 3 years after study enrollment
Population: Only eligible patients are considered in the analysis of this outcome measure
Measure: Number (95% Confidence Interval); unit: Percent Probability
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 37 | 37
Percent Probability | 94.59 [80.07 to 98.62] | 91.74 [76.52 to 97.26]

5. Secondary Outcome: Number of Patients With Toxic Events After 2 Dose Reductions
Description: Number of patients who have an additional significant toxicity coded using Common Terminology Criteria for Adverse Events Version 5.0 after experiencing two dose reductions from their assigned treatment dose.
Time Frame: While receiving protocol therapy up to 3 years after study enrollment
Population: Only eligible patients are considered in the analysis of this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 37 | 37
Participants | 2 | 16

6. Secondary Outcome: Pharmacokinetic Parameters of Lenalidomide
Description: Concentration of lenalidomide obtained from any day between day 5 and 21 of the first cycle of chemotherapy in nanograms per mL.
Time Frame: Between days 5-21 of course 1 and each dose reduction
Population: Only eligible patients who have lenalidomide concentration measure are considered in the analysis of this secondary outcome measure
Measure: Median (Inter-Quartile Range); unit: nanograms per mL
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 22 | 25
nanograms per mL | 15.1 [7.0 to 36.8] | 178.8 [68.5 to 391.7]

7. Secondary Outcome: Magnetic Resonance Imaging Sequence
Description: Response categories (complete response, partial response, stable disease, and progression) will be determined from the following three standard magnetic resonance sequences, T2-weighted, fluid attenuated inversion recovery, T1-weighted post-contrast. Percent agreement between the sequences will be estimated as the number of follow-up scans in which the corresponding sequence agreed divided by the total number of follow-up scans.
Time Frame: Up to 3 years
Population: Scans completed and reviewed by standard magnetic resonance sequences. Only eligible patients are considered in the analysis of this outcome measure.
Measure: Number; unit: Number of scans in agreement
Units Other Than Participants: Scans
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
Number analyzed (Participants) | 30 | 25
Number analyzed (Scans) | 110 | 77
Number of scans in agreement
  T1-weighted post-contrast and fluid attenuated inversion recovery: number analyzed (Participants) | 25 | 23
  T1-weighted post-contrast and fluid attenuated inversion recovery: number analyzed (Scans) | 64 | 63
  T1-weighted post-contrast and fluid attenuated inversion recovery | 35 | 43
  T1-weighted post-contrast and T2-weighted: number analyzed (Participants) | 25 | 23
  T1-weighted post-contrast and T2-weighted: number analyzed (Scans) | 64 | 63
  T1-weighted post-contrast and T2-weighted | 35 | 42
  Fluid attenuated inversion recovery and T2-weighted: number analyzed (Participants) | 29 | 25
  Fluid attenuated inversion recovery and T2-weighted: number analyzed (Scans) | 108 | 77
  Fluid attenuated inversion recovery and T2-weighted | 66 | 60

ADVERSE EVENTS:
Time Frame: AEs and OAEs: Up to 6 months post-treatment planned as 3 years; All-Cause Mortality: up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Arm I (Low-dose Lenalidomide) | Arm II (High-dose Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 4/37 | 4/37
Serious Adverse Events (participants affected / at risk) | 6/37 | 16/37
Other Adverse Events (participants affected / at risk) | 15/37 | 30/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose Lenalidomide) (N=37) | Arm II (High-dose Lenalidomide) (N=37)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2) | 5 (5)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphasia (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Hydrocephalus (Nervous system disorders) | 4 (4) | 2 (2)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 3 (3)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Low-dose Lenalidomide) (N=37) | Arm II (High-dose Lenalidomide) (N=37)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 4 (4)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4) | 4 (4)
Neutrophil count decreased (Investigations) | 9 (9) | 21 (21)
Platelet count decreased (Investigations) | 0 (0) | 6 (6)
Weight gain (Investigations) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 1 (1) | 11 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT01553149/Prot_SAP_001.pdf